CLINICAL TRIAL: NCT02318745
Title: Preventing Health Disparities in Hispanic Youth
Acronym: CIFFTA-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daniel A. Santisteban, Ph.D., Clinical Psychologist/Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20070334; P60MD002266 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: ADHD; Conduct Disorder; Depression; Family Dysfunction
Keywords: Family Therapy; Substance abuse prevention; Minority; randomized trials; outcome research; adolescent treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally Informed Family Treatment for Adolescents (Experimental): CIFTA focuses on improving parenting practices, parent-adolescent attachment, adolescent ability to meet developmental challenges, increasing family support and decreasing family conflict/negativity, increasing knowledge of drug effects and triggers to use. Parents are taught general parenting and how to help a son or daughter with depression, conduct problems, and/or ADHD. Psycho-educational modules complement the family therapy and culturally relevant information is infused throughout the treatment. In family therapy sessions family members practice the skills and psycho-educational material they have learned. Treatment last approximately 4 months and includes approximately 6 session per month. Session may be family therapy sessions, individual sessions, or psycho-educational modules.
  Interventions: Behavioral: Culturally Informed Family Treatment for Adolescents
- Individual Treatment As Usual (Active Comparator): The active comparison condition reflects the typical individually-oriented services that behavior problem youth receive in the community. It was designed to isolate the effects of the CIFTA family interventions. A community agency helped us to standardize the individually-oriented services that were normally provided and a therapist trained by that agency was hired to work on the study to provide continuity to the services. The adolescent individual sessions addressed depression, ADHD, and/or conduct disorder through Cognitive Behavior Therapy, Interpersonal psychotherapy, social skills training, anger control training, problem solving skills, and assertiveness training. The ITAU therapists were expected to hold 6 sessions per month with the youth.
  Interventions: Behavioral: Individual Treatment

INTERVENTIONS:
Behavioral: Culturally Informed Family Treatment for Adolescents — Family Therapy, Psycho-educational Modules, Individual therapy sessions
  Arms: Culturally Informed Family Treatment for Adolescents
Behavioral: Individual Treatment — Cognitive Behavior Therapy, Interpersonal psychotherapy, social skills training, anger control training, problem solving skills, assertiveness training, and the Empty chair technique from Gestalt therapy
  Arms: Individual Treatment As Usual

SUMMARY:
This study seeks to investigate the efficacy and mechanisms of a highly promising "Culturally Informed Family Therapy for Adolescents" in preventing the emergence of two important health disparities in Hispanic youth, namely drug use & HIV and other sexually transmitted infections (STI). The proposed study is submitted as part of a P60 application entitled "NCMHD Center for Culturally-Tailored Hispanic Health Disparities Research (El Centro)", in response to the NIH RFA-MD-06-002: Establishing Comprehensive NCMHD Research Centers of Excellence.

This study investigates: 1) the efficacy of the treatment in reducing existing psychiatric, behavioral and family problems in youth, and 2) the indicated prevention effects of the intervention on the emergence of drug use and HIV/STI 20 months after baseline. There is a substantial literature linking disruptive behaviors (i.e., conduct disorder and attention deficit hyperactivity disorder) and mood instability (i.e., depressive disorders) and family conflict to the development of the Hispanic health disparities of drug use and HIV/STI. Conduct disorder (CD), attention deficit hyperactivity disorder (ADHD) and depressive disorders (DD) will be targets of treatment, as will be the family risk factors (e.g., poor parenting, family conflict) and acculturation-related stressors, all of which have been shown to place youth on a destructive trajectory toward deteriorating health.

DETAILED DESCRIPTION:
DESIGN AND METHODS. Overview. The first phase of the proposed study will include minor adaptations to the manual to enhance its "fit" with the specific characteristics of the target population, finalizing all assessment measures, finalizing the list of CTAU agencies and the referral mechanisms, conducting therapist training for the CIFTA conditions and assessor/interviewer training, and strengthening our connections with referral sources (months 1- 5). The team is experienced in all of these activities from previous treatment development and clinical trial projects. Immediately following this phase, the investigators will begin to recruit adolescents (11-14 years of age) who meet DSM-IV criteria for two of the following diagnoses (CD, DD, ADD) OR DSM-IV criteria for one diagnosis (CD, DD, ADD) and severe family conflict. Following screening, consent and assessment, the adolescents and their families will be randomly assigned to either the (1) Community Treatment as Usual Agency, or the (2) Culturally Informed Family Therapy for Adolescents. Assessments will be conducted at baseline (T1), post-treatment (T2- 4 months), follow-up 1 (T3- 12 months post baseline) and follow-up 2 (T4- 20 months post baseline). Data from service utilization and self-reports of therapeutic alliance will also be collected throughout the entire course of therapy. Longitudinal data analysis (growth curve modeling) will be used to test study hypotheses. Each of the specific components and procedures are described in detail below.

Design for Manualization of Refinements. The investigators and clinical team have experience in manualizing key treatment components. Although relatively minor, some of the specific refinements the investigators propose, based on our prior experience with CIFTA will include: 1) revising the parent training modules to be developmentally appropriate to middle school ages, 2) the establishment of healthy social activities that can shape the selection of prosocial peer groups and activities before ties to deviant peers are crystallized, 3) the creation of family session material that facilitates the parent-child discussion of country and culture of origin and helps to explore questions about the child's ethnic identity.

Manual Refinement meetings will include counselors and investigators and will be held to clarify the precise nature of the new material to be delivered, the therapeutic processes and procedures that are optimal for delivery of the material, and the interaction between these interventions and other intervention components. New manual entries/clarifications will be written together during the meeting so that the language is recommended and approved by both clinicians and investigators. The investigators have utilized this method in all of our treatment development efforts and the investigators have found that it leads to language that is user-friendly for clinicians. The team also agrees on adherence checklist items that reflect the nature of the intervention.

Therapist Selection, Training and Supervision. Two therapists (.3 FTE each) will deliver the CIFTA intervention. These therapists will be primarily selected from the Center for Family Studies, which has a cadre of therapists that have extensive experience with Hispanic youngsters and have had experience in delivering manualized treatments within a clinical research context. All therapists must also have at least a master's degree in counseling, psychology, social work or a related field. Therapists selected for this study must be bilingual (Spanish and English) to ensure that primarily Spanish-speaking family members can fully participate.

Therapist training. Training will follow the format the investigators have used over many years and also currently utilize in our Training Institute. The first phase of training will consist of a 3-day training workshop that includes the use of didactic material, the treatment manuals, and the presentation of videotaped sessions from our pilot work. The second phase will include intervention implementation with 1 pilot case. A therapist will be required to work with a pilot case for at least a one-month to be certified in that condition. The guidelines for certification the investigators will use are similar to those proposed by Carroll (1998) and will focus on the implementation of key aspects of the revised CIFTA treatment (parenting, skills modules, cultural modules, etc). Key aspects of therapy that receive poor ratings will require retraining. Interventions will be delivered over one month, a briefer period than is typical of the actual intervention in the trial, but will be sufficient to ensure comfort and competence in the key treatment components. There will be a 2 day workshop following the pilot phase to solidify any issues that remain and to incorporate any manual clarification that will assist in achieving high levels of competence and fidelity/adherence. The PI has extensive experience as a workshop trainer in family-oriented and substance abuse interventions.

Therapist Supervision and Adherence Monitoring. Weekly clinical meetings will be held for the CIFTA therapists. Dr. Santisteban will supervise the team and provide formal supervision to all project team members. All sessions will be videotaped and these will be reviewed. The clinical complexity of cases will be discussed and good culturally-competent and clinical implementation will be emphasized.

Adherence raters will be trained using the established adherence checklists for the two study conditions. The condition supervisor will be held as the gold-standard for inter-rater reliability on adherence ratings and raters will be trained to achieve an intra-class correlation coefficient of .70 or higher, and at least 80% agreement across items. Inter-rater reliability will be checked regularly to avoid drift. Specifically, an independent adherence rater will randomly select 10% of the video-taped sessions from each condition at different treatment phases (early, mid, and late) for adherence ratings. These ratings will document the adequacy with which treatment sessions follow specific manual interventions and treatment strategies. Ratings that fall below adequacy on any dimension/component will trigger increased supervision focused for that dimension and if necessary, re-training.

Participants for the randomized trial. 200 11-14 year old Hispanic youngsters meeting DSM-IV criteria for multiple child disorders (including CD, ADHD, and DD [any of the depressive disorders}) will be included in the study along with their families. Participants will be recruited from the community in general as well as from the Dade County Public School System, the University of Miami Institute for Individual and Family Counseling, and MBHC/Spectrum Programs. The investigators will work intensively with referral sources to ensure full representation of both males and females (goal will be to obtain 50%/50% split in boys and girls) and a diverse mix of Hispanic subgroups that are prominent in the South Florida area (e.g., Mexican, Central American, South American, Puerto Rican, and Cuban). Randomization will be stratified by gender, symptom profile, and years residing in U.S.

Participants will go through a screening to evaluate if they meet criteria for the study and then will complete baseline (T1) and randomization. Assessments will be conducted again at post-treatment (T2- 4 months), follow-up 1 (T3- 12 months post baseline) and follow-up 2 (T4- 20 months post baseline). The 4, 12 and 20 month assessments have been selected to coincide with the termination of treatment, follow-up 12 months after baseline, and 20 months after baseline.

Participant Recruitment Plan. The Center for Family Studies has fostered a collegial and continuous relationship with many of the referral sources in the community. Given this relationship, in our last studies the investigators surpassed the number of participants originally proposed. In addition, the investigators have had experience recruiting and assessing youth from these sources (Santisteban, Coatsworth, et al., 1997; Santisteban, Dillon, et al., 2005). The main referral sources for our proposed study will be the community in general as well as the Dade County Public School Sytem, the University of Miami Institute for Individual and Family Counseling and MBHC/Spectrum Programs. These clinics are very active, with a large percentage of Hispanic families and fully capable of referring a large number of cases per week (only approximately 5 cases per month are needed). The investigators have strong referral relationships with the Dade County school system counselors who referred the large majority of the cases for the Santisteban et al. (1997) study which was a precursor to the current study, and with the Miami Behavioral Health Center which is the main agency treating mental health issues in the Hispanic population. Because our Center has a history of leadership on Hispanic issues, the investigators are looked upon for culturally competent treatment of youth and families.

Throughout the study the investigators plan to conduct meetings in the schools with the school counselors and at the Institute for Individual and Family Counseling Clinic with the therapists to explain the specifics of this new study. Throughout the life of the study, the assessors will participate in the staffing meetings to consult with staff as needed at the Insititute for Individual and Family Counseling on a weekly basis, as well as maintain weekly contacts with school counselors to obtain referrals. We will encourage counselors from the schools and clinicians from the Institute for Individual and Family Counseling Clinic to call the Study Assessor in the presence of the family, once they have introduced the study to the family and they expressed interest in the study. The assessor will then make an appointment with the family for study consent and initial screening. In the case the assessor is not available, the counselors will ask for the family's permission to give the assessor their phone number to be contacted at a later time. The same process will be used at MBHC/Spectrum Programs. As mentioned before, this referral process has been very successful in past studies; thus we anticipate similar success in the proposed study. We will also meet with individuals involved with the media and radio and any other community referral source that would be appropriate as a referral source. In addition, we have created a brochure with important information about the research study to be given to referral agencies/sites via e-mail and/or in person and for potential participants. We will also run ads in several community based newspaper in order to assist in the recruitment of participants.

Inclusion criteria. To be included in the study, the youngster/families must meet the following criteria: (a) be between the ages of 11 to 14 years old, (b) be born in a Spanish speaking country or have parents born in Spanish speaking countries, (c) be living with at least one family member of an older generation such as a parent or grandparent; and all family members of the household (including the youngster and at least one adult) must agree to be present during the assessment and treatment sessions, and (d) meet DSM IV criteria for two of the following diagnoses (CD, DD, ADD) OR DSM-IV criteria for one diagnosis (CD, DD, ADD) and severe family conflict.

Exclusion criteria. Participants who meet any of the following will be excluded: (a) history of any of the following DSM IV diagnoses - Pervasive Developmental Disorders, Elective Mutism, Organic Mental Disorders (except Psychoactive Substance-Induced), Schizophrenia, Delusional (Paranoid) Disorder, Psychotic Disorder, and Bipolar Affective Disorder, (b) Any Substance Abuse or Dependence Disorder diagnosis (substance use that does not meet DSM IV diagnosis criteria will not excluded).

Inclusion of family members in the study. Youth and both parents are scheduled for assessment. All family members living in the household of the target adolescent will be invited to participate. Decisions are made on a case by case basis regarding the inclusion of very young children (younger than 10). In addition, individuals who are not blood relatives but have significant roles in raising the adolescent will also be invited. Parental figures will be asked to complete the parent version of the assessment battery. Our previous projects have been very successful at identifying and engaging family members into treatment as well as in retaining them throughout the course of the treatment (Santisteban et al., 1996; Szapocznik et al., 1988).

Screening and Assessment Procedures. Families that are interested will have the research study explained to them, and will be asked to sign an informed consent that explains the study. Research assessors will be trained to conduct the initial screening using the Diagnostic Interview Schedule for Children (DISC) and the Family Environment Scale - Conflict Scale. All participants included in the study will complete a Baseline assessment and will be randomized after testing. Assessments will be conducted again at post-treatment (T2- 4 months), follow-up 1 (T3- 12 months post baseline) and follow-up 2 (T4- 20 months post baseline). A trained Master's-level research assistant who is bilingual in English and Spanish will administer all assessments. Our assessors have worked on multiple projects using the self-reports and interview measures proposed in this study. All measures and consents will be available in Spanish to ensure that primarily Spanish-speaking adolescents or parents are not excluded.

Each assessment interview will last approximately 3 hours and consist of three components: an individual interview with the adolescent, an individual interview with each parent/guardian, and a family interview session.

Prevention of Dropouts from the study. To ensure capturing and maintaining as much of the sample as possible, each participant will have contact with the same assessment specialist during the entire course of the study. Having the same assessor follow a given family throughout the study will provide personal continuity, and thus improve participation and retention in the study. Additional procedures that we have established to retain participants in prior studies, and ensure follow-up assessments, include: 1) conducting assessments at convenient locations for the families including their homes when necessary, 2) providing compensation to families for their participation in assessments, 3) conducting the service utilization phone interviews at baseline and 4, 8, 12, 16, and 20 months post-baseline, 4) updating all contact information at regular intervals, 5) obtaining the names of three contact persons who are close to family members and who may be contacted by the Assessment Specialist in the event that the family is unreachable at the assessment time-points (this is included in the consent form), and 6) sending out birthday and holiday cards to all participants. In our experience, the utilization of standard operating procedures for tracking and contacting participants dramatically increase retention rates in the study. The PI and research team has solid experience with tracking families for follow-up related activities. In our last federally funded treatment development grant we were able to track families six weeks after the adolescent was discharged from an Addictions Receiving Facility at a success rate of 96%.

AIM I: To refine/adapt the CIFTA treatment manual to meet the unique clinical and developmental characteristics of youth 11-14 years of age, while at the same time targeting existing psychiatric, behavioral and family problems (CD, ADHD, DD, family dysfunction) via a "flexible" treatment manual that can tailor the intervention package to youth and their families.

AIM II: To test, using a randomized clinical trial, the efficacy of CIFTA compared to a Community Treatment-as-Usual (CTAU) in reducing symptoms of CD, ADHD, DD, and family dysfunction.

AIM III: To test the ability of CIFTA, compared to CTAU, to prevent health disparities conditions (drug use andHIV/STI) over a period of 20 months post baseline.

AIM IV: To empirically (using cluster analysis) identify subtypes of profiles on acculturation and immigration-related factors, and to investigate the relationship of these culture-related subtypes to problem behavior profiles and to responses to the CIFTA treatment.

AIM V: To investigate the relationship of CIFTA's hypothesized mechanisms of treatment change (parenting practices, parent-school interactions, child utilization of skills, etc) to CIFTA treatment outcome on the existing problems (CD, ADHD, DD, family dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* 11-14 year old Hispanic youngsters meeting DISC-Predictives cut-off scores for two or more disorders (including CD, ADHD, and
* DD [any of the depressive disorders]) and/or family conflict were included in the study along with their families.

Exclusion Criteria:

* Participants who meet any of the following will be excluded:

  * History of any of the following DSM IV diagnoses - Developmental Disorders, Elective Mutism, Organic Mental Disorders (except Psychoactive Substance-Induced), Schizophrenia, Delusional (Paranoid) Disorder, Psychotic Disorder, and Bipolar Affective Disorder,
  * Any Substance Abuse or Dependence Disorder diagnosis (substance use that does not meet DSM IV diagnosis criteria will not excluded).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  The Child Behavior Checklist (CBCL; Achenbach, 1991) was used as the parent report of youth's problem behaviors. Problem behaviors were scored along the dimensions of the super-ordinate domains of "internalizing" and "externalizing" behaviors. Smaller syndromes of behavior problems (e.g. delinquent behavior, aggressive behavior, anxious/depressed) were also available. The two syndromes that comprise the externalizing dimension, delinquent behavior and aggressive behavior were used as indicators of behavior problems, whereas the anxious/depressed dimension was used as an indicator of internalizing problems. Internal consistency reliabilities of each of the subscales ranged from .73 to .90.
Youth Self Report Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  The Youth Self-Report (YSR; Achenbach, 1991) was used as the adolescent (11-18 years old) self-report instrument to assess problem behaviors, and the degree of functioning on three dimensions of Social Competence. Problem behaviors were scored along the dimensions of the super-ordinate domains of "internalizing" and "externalizing" behaviors. As with the CBCL, smaller syndromes of behavior problems (e.g. delinquent behavior, aggressive behavior, anxious/depressed) were also available. The two syndromes that comprised the externalizing dimension, delinquent behavior and aggressive behavior were used as indicators of behavior problems, whereas the anxious/depressed dimension was used as an indicator of internalizing problems. Internal consistency reliabilities of each of the subscales ranged from .72 to .90.
Diagnostic Interview Schedule for Children - Predictives Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  The Diagnostic Interview Schedule for Children - Predictive Scales (DISC-P; Lucas et al., 1997) was used to evaluate psychiatric symptoms in a standardized manner consistent with DSM diagnostic criteria. For this study, the Attention Deficit Hyperactivity Disorder, Depression, Oppositional Defiant Disorder, and Conduct Disorder components of the measure were used. The DISC-P has been found to have a high degree of sensitivity with respect to the DISC for specific DPS scales. The DISC-P was administered to both parents and children.
Substance Use and Attitudes Regarding Substance Use Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  We combined items from several instruments. Items extracted from the Monitoring the Future Study (Johnston, O'Malley, & Bachman, 2003) asked whether or not the adolescent had used cigarettes, alcohol, and other illegal substances. Adolescents who responded to using an illegal substance were asked to respond to the type of substance used, age of first use, and the frequency of use in the past 30 days. Items from the CSAP National Student Survey (1996), and the USC Health Behaviors Survey (Pentz, et al., 1989) measured attitudes toward tobacco, alcohol, and illegal substances, intentions regarding substance use, the degree to which adolescents care about how others would view them if they used drugs or alcohol, and perceptions of parents, peers, teachers approval/ disapproval of respondent's tobacco, alcohol, or other drug use. High internal consistency for the attitudes, intentions, and social norms subscales have been found (.92, .99, and .97, respectively).
Adolescent Risky Sexual Behaviors Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  Questions from several instruments were combined into one gated instrument to assess a range of sexual risky situations and behaviors in the youth. Some questions from the Interview on Situations of Sexual Possibility- Booklet A (ISSP; Paikoff, 1995), a gated, structured interview about unsupervised peer activities, situations of sexual possibility, and other questions from the Sexual Behavior instrument (Jemmot, Jemmot, & Fong, 1998), that assess the adolescent's sexual behavior, condom use, and existence of a sexually transmitted disease during their lifetime and in the past three months were combined. There was a total of 19 items in the questionnaire, however, the instrument is gated and not all questions were asked. Depending on the types of risky situations the adolescent had been involved in, the questions become more specific about risky sexual involvement or the instrument was discontinued if the adolescent had not been exposed to certain behaviors.

SECONDARY OUTCOMES:
Family Environment Scales Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  The Cohesion and Conflict scales from the FES (Moos & Moos, 1994) were be used in this study. The Cohesion scale measured the extent to which the adolescent or parent views the family as harmonious and close. The Conflict scale measured the extent to which the adolescent or parent views the family as characterized by frequent disagreements. These two constructs have been found to be among the strongest family-based correlates of adolescent problem behavior. Moreover, these two scales (18 items) have been used successfully in previous research conducted by the investigator on adolescent treatment outcomes (Santisteban, Coatsworth, et al., 2003). Internal consistencies based on data from a normative sample for the cohesion and conflict scales were .78 and .75, respectively. Parents and youth completed this questionnaire and internal consistency reliabilities ranged from .67 to .76 for the parents and from .75 to .76 for the youth.
Parenting Practices Questionnaire Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  Parenting Practices Questionnaire (PPQ). The Parenting Practices Questionnaire (Gorman-Smith et al., 1995) from the Chicago Youth Development Study was used to assess four dimensions of parenting behavior: Positive Parenting, Discipline effectiveness, Discipline Avoidance and Extent of Involvement. Positive parenting and extent of involvement were assessed only in the adolescents. Internal consistency reliabilities of each of the subscales ranged from .64 to .80 in the parents and .76 to .87 in the adolescents.
Parental Monitoring Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  Parental Monitoring Instrument. The PMI (Cottrell et.al. 2007) was developed to determine how often parents use seven monitoring strategies: direct monitoring, indirect monitoring, school, health, computer, phone, and restrictive. The scale contains 27 items with 4 frequency responses (0 times, 1 to 2 times, 3 to 4 times, and 5-plus times). Parents and adolescents reported how many times parents used a specific monitoring strategy in the past 4 months. Internal consistency reliabilities were .88 and .83 for the parents and youth, respectively.
Parent Child Attachment Change Measure | Baseline, T2 (4 months post baseline), T3 (12 months post baseline), and T4 (20 months post baseline)
  Parent-Adolescent Attachment. The Inventory of Parent and Peer Attachment (IPPA) (Armsden & Greenberg, 1987) was used to assess adolescents' perception of the positive and negative aspects of their attachment to their parents. The IPPA measures three dimensions: degree of mutual trust, quality of communication, and the extent of alienation. Internal consistency reliabilities of each of the subscales ranged from .76 to .91.